CLINICAL TRIAL: NCT00220948
Title: Large Array EMG Discriminability in Discogenic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Texas Back Institute (Other)
Collaborators: CERSR (Unknown); Innovative Spinal Technologies, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: P699
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2005-09-22 (Estimated); Status verified 2005-07

CONDITIONS: Discogenic Pain
Keywords: discogenic pain; myoelectric activity

INTERVENTIONS:
Procedure: CERSR Myoelectric monitoring during standardized tasks

SUMMARY:
Hypothesis:

Myoelectric patterns observed from the CERSR array during standardized testing are sensitive in identifying healthy subjects from patients with internal disc derangement and a positive discogram. A positive CT discogram is defined as one following the Dallas discogram protocol with abnormal disc morphology and reproduction of symptoms

DETAILED DESCRIPTION:
Methodology:Patient Inclusion / Exclusion Criteria:Patient's who present with non-radicular low back with or without sclerotomal, referred leg pain and who have failed conservative care for 5 months or otherwise meet clinical criteria for performing diagnostic discography are potential candidates for recruitment in this study. The criteria are as follows:Inclusion / Exclusion:· Age 21 - 55· No prior spine surgery.· No neurological deficit.· VAS > 3.0· The patient has been referred for provocative discogram diagnostic study with a suspected single level internal disc derangement.· Normal psychometric screening.For healthy control subjects the criteria will be as follows:· Age 21 - 55· No spinal deformity· No prior spine surgery.· No history of disabling back or leg pain.· No history of back pain for the past 6 months year. Patient Recruitment: A total of 80 subjects, divided into four groups ( 20 per group), are being sought for this study. Group C will be a population of healthy control subjects to be compared with Group U, unhealthy subjects. Group U will represent the first 20 patient participants who are referred for discogram procedures. Group DP will consist of a separate group of 20 patients being referred for discogram testing whose results are positive. Group DN will consist of 20 patients whose discogram results are negative. Statistical criteria for valid analysis requires separate non-overlapping grouping of patients to maintain the accuracy of the Type 1 error estimate in the analysis of results. A total of 80 patients will be sought as the analysis of sensitivity and specificity requires a minimum number of false positive and false negative results to be present in each subgroup for the analysis to be performed. The TBI practice is equipped with electronic scheduling, medical record and billing systems. This poses significant advantages for patient recruitment to this project. On a daily basis, the Project Coordinator (PC) can access daily schedules for patients entering the system for all 17 TBI physicians. This can be cross-correlated later with exiting diagnosis and diagnostic orders to ensure maximum capture of potential candidates.The attending physician's medical assistant, on being notified of the need for a discogram, will contact the PC. The PC then will review the chart and confer with the attending provider to confirm entrance requirements. The patient will be asked for permission to be contacted by the PC for soliciting participation in the project. Upon obtaining permission, the PC will contact the patient and explain the project and signed informed consent obtained from those who agree to participate. Those whom do not sign consent to participate or consent to be monitored will continue with their care and be purged from the project records. Patients will then be scheduled for CERSR evaluation prior to performance of the diagnostic procedure. The PC will perform the CERSR test at the designated appointment and will provide the Principal Investigator (PI) with the test results for interpretation without identification of which diagnostic procedure or group assignment the patient is in. To ensure blinding of the PI, the demographic fields usually maintained in the CERSR software will be left blank with the exception of the patient identifier. Separate records will be maintained by the PC with respect to this information as well as report of findings from discogram as may be appropriates.The surgeon co-investigator will review the discogram results on each patient and partition them into positive and negative results based both on morphologic and pain concordance criteria. Testing will continue until a full block of 20 subjects for each group is obtained. The PC will also solicit healthy subjects from the TBI and Presbyterian Hospital staffs numbering several hundred in total. All healthy volunteers will be compensated $50.00 for their time and inconvenience in participation in the CERSR test. Psychometric Screening: Psychometric screening of all participants (healthy and patient) will be performed using the SCL90-R. This instrument has been used successfully for years as a strong psychometric screening tool that incorporates evaluation for somatization. Our consulting psychologist, Dr. Block, whose sole practice for 15 years has been the evaluation and treatment of spine pain patients, will perform the scoring of the SCL90-R. Subjects whose scores are high on the somatization scale alone or whose total scores are suggestive of strong psychosocial component will not be included.CERSR Evaluation and Interpretation:The CERSR evaluation will consist of the standardized tests for upright standing, flexion and weight bearing. Interpretation will similarly follow the proscribed method considering the maximum RMS, uniformity, centrality, organization and location as described in the Appendix I. Outcome of the analysis will the classification of the patient into disc, healthy or other.. Interpreter blinding:The PI will perform interpretation of the CERSR tests without knowledge of the patient's group membership. The surgeon co-investigator will assess discogram results without knowledge of the CERSR test results. At the end of the study, PI interpretation will be joined with the database on subject status and patient outcome from diagnostic testing, as appropriate. Analysis will be performed with patients grouped according to their group status (C, U, DP, DN).Interpretation of Diagnostic Testing:A positive discogram will be determined following the Dallas protocol for abnormal morphology within the inner disc and the reproduction of exact pain or similar pain with disc pressurization.AnalysisAnalysis 1: Healthy (n=20) Unhealthy (n=20) Abormal CERSR False Positive Positive Normal CERSR Negative False Negative Analysis 2: Disco Positive(n = 20) Disco Negative(n = 20) Abnormal CERSR Positive False Positive Normal CERSR False Negative Negative Using the proprietary CERSR methods of analysis (max RMS, uniformity, centrality, organization) to classify patients into healthy, disc or other. Sensitivity, specificity and predictive values will be calculated for patients who are healthy versus those who have positive and negative CERSR tests. This analysis will establish the minimum boundaries of the CERSR technology and its ability to differentiate normal from unhealthy subjects as well as establish the generalizability of interpretation in the hands of this investigative group. A healthy subject whose CERSR test is identified as having characteristics of unhealthy patients will be classified as a false positive. Patients with suspected discogenic pain who fail to be classified by myoelectric patterns as unhealthy will be identified as having false negative tests. The second analysis will examine sensitivity, specificity and predictive values for differentiating discogenic pain generators from non-discogenic pain generators. Patients with positive CERSR tests for disc patterns of pain who are classified by discogram as being negative will be considered false positives. Patients with negative CERSR tests who are classified by discogram as being positive for discogenic pain will be considered false negatives. This test will distinguish the accuracy of pattern in separating discogenic pain from nondiscogenic sources.

ELIGIBILITY:
Inclusion Criteria:

Patients: Failed conservative care > 5 months, Age 21 - 55.VAS > 3.0· The patient has been referred for provocative discogram diagnostic study with a suspected single level internal disc derangement.· Normal psychometric screening.

Healthy Subjects: · Age 21 - 55

Exclusion Criteria:

* Prior spine surgery.Neurological deficit.·Spinal deformity· Prior spine surgery.·History of disabling back or leg pain.·

Healthy subjects: History of back pain for the past 6 months year.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60
Dates: Start 2004-08; Study Completion 2006-03

PRIMARY OUTCOMES:
Agreement between discogram interpretation and myoelectric interpretation

CONTACTS AND LOCATIONS:
Overall Officials: John J Triano, DC,PhD, Principal Investigator — Texas Back Institute and University of Texas, Arlington
Locations (1):
- Texas Back Institute, Plano, Texas, United States